CLINICAL TRIAL: NCT01826929
Title: Effectiveness of a New Health Care Organization Model in Primary Care for Chronic Cardiovascular Disease Patients Based on a Multifactorial Intervention: The PROPRESE Randomized Controlled Trial.
Brief Title: Effectiveness New Health Care Organization Model in Primary Care for Chronic Cardiovascular Disease Patients Based
Acronym: PROPRESE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: USI-10-66; SM I 14/2010 (Other Grant/Funding Number: Valencia Regional Ministry of Health)
Record Dates: First submitted 2013-03-25; First posted 2013-04-09 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Ischemic Heart Disease
Keywords: Health Services Research; Cardiovascular Diseases; Primary Care; Secondary Prevention.
MeSH Terms: conditions — Myocardial Ischemia; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic education (Experimental): Organized intervention strategy:Informed active patient, shared decision making, appointment planning, primary care doctor-nurse teamwork, actions based on scientific evidence.
  Interventions: Other: Therapeutic education
- Usual care model (No Intervention)

INTERVENTIONS:
Other: Therapeutic education
  Arms: Therapeutic education

SUMMARY:
The purpose of this study is to determine whether a multifactorial primary care intervention based on chronic models can improve the level of control and reduce the number of hospital admissions in patients with ischemic heart disease.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of IHD of any site (ICD-10 codes from 410 to 414 inclusive.
* signed written informed consent

Exclusion Criteria:

* lack of consent
* immobilized patients
* patients with serious health problems or with a low life expectancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Number of hospitalizations/cause at 12 months | Baseline and 12 months

SECONDARY OUTCOMES:
Change from baseline Blood pressure | Baseline, 4 months, 8 months and 12 months.
  It is measured at each visit in order to monitor the evolution. However, the change is calculated as the latest time point minus the earliest time point.
Change from baseline LDL cholesterol | Baseline, 4 months, 8 months and 12 months.
  It is measured at each visit in order to monitor the evolution. However, the change is calculated as the latest time point minus the earliest time point.
Change from baseline Body Mass Index | Baseline, 4 months, 8 months and 12 months
  It is measured at each visit in order to monitor the evolution. However, the change is calculated as the latest time point minus the earliest time point.
Change from baseline Basal Blood Glucose | Baseline, 4 months, 8 months and 12 months
  It is measured at each visit in order to monitor the evolution. However, the change is calculated as the latest time point minus the earliest time point.
Change from baseline Healthy Life Habits (exercise, mediterranean diet) | Baseline, 4 months, 8 months and 12 months
  It is measured at each visit in order to monitor the evolution. However, the change is calculated as the latest time point minus the earliest time point.
Change from baseline Number of annual primary care visits | Baseline and 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Sant Joan d'Alacant, Alicante
  - Castellon, Castellon
  - Valencia, Valencia

REFERENCES:
- [Background] Lorig KR, Ritter PL, Dost A, Plant K, Laurent DD, McNeil I. The Expert Patients Programme online, a 1-year study of an Internet-based self-management programme for people with long-term conditions. Chronic Illn. 2008 Dec;4(4):247-56. doi: 10.1177/1742395308098886. PMID 19091933
- [Background] Banegas JR, Rodriguez-Artalejo F, Graciani A, Villar F, Herruzo R. Mortality attributable to cardiovascular risk factors in Spain. Eur J Clin Nutr. 2003 Sep;57 Suppl 1:S18-21. doi: 10.1038/sj.ejcn.1601804. PMID 12947446
- [Background] Graham I, Atar D, Borch-Johnsen K, Boysen G, Burell G, Cifkova R, Dallongeville J, De Backer G, Ebrahim S, Gjelsvik B, Herrmann-Lingen C, Hoes A, Humphries S, Knapton M, Perk J, Priori SG, Pyorala K, Reiner Z, Ruilope L, Sans-Menendez S, Scholte op Reimer W, Weissberg P, Wood D, Yarnell J, Zamorano JL, Walma E, Fitzgerald T, Cooney MT, Dudina A; European Society of Cardiology (ESC) Committee for Practice Guidelines (CPG). European guidelines on cardiovascular disease prevention in clinical practice: executive summary: Fourth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (Constituted by representatives of nine societies and by invited experts). Eur Heart J. 2007 Oct;28(19):2375-414. doi: 10.1093/eurheartj/ehm316. Epub 2007 Aug 28. No abstract available. PMID 17726041
- [Background] Lobos JM, Royo-Bordonada MA, Brotons C, Alvarez-Sala L, Armario P, Maiques A, Mauricio D, Sans S, Villar F, Lizcano A, Gil-Nunez A, de Alvaro F, Conthe P, Luengo E, Del Rio A, Cortes O, de Santiago A, Varga MA, Martinez M, Lizarbe V; Comite Espanol Interdisciplinario para la Prevencion Cardiovascular. [European Guidelines on Cardiovascular Disease Prevention in Clinical Practice. CEIPC 2008 Spanish adaptation]. Rev Clin Esp. 2009 Jun;209(6):279-302. Spanish. PMID 19635253
- [Background] Selby JV, Schmittdiel JA, Fireman B, Jaffe M, Ransom LJ, Dyer W, Uratsu CS, Reed ME, Kerr EA, Hsu J. Improving treatment intensification to reduce cardiovascular disease risk: a cluster randomized trial. BMC Health Serv Res. 2012 Jul 2;12:183. doi: 10.1186/1472-6963-12-183. PMID 22747998
- [Background] Kotseva K, Wood D, De Backer G, De Bacquer D, Pyorala K, Keil U; EUROASPIRE Study Group. Cardiovascular prevention guidelines in daily practice: a comparison of EUROASPIRE I, II, and III surveys in eight European countries. Lancet. 2009 Mar 14;373(9667):929-40. doi: 10.1016/S0140-6736(09)60330-5. PMID 19286092
- [Background] Brotons C, Permanyer G, Pacheco V, Moral I, Ribera A, Cascant P, Pinar J; PREMISE study group. Prophylactic treatment after myocardial infarction in primary care: how far can we go? Fam Pract. 2003 Feb;20(1):32-5. doi: 10.1093/fampra/20.1.32. PMID 12509367
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness: the chronic care model, Part 2. JAMA. 2002 Oct 16;288(15):1909-14. doi: 10.1001/jama.288.15.1909. PMID 12377092
- [Background] Davino-Ramaya C, Krause LK, Robbins CW, Harris JS, Koster M, Chan W, Tom GI. Transparency matters: Kaiser Permanente's National Guideline Program methodological processes. Perm J. 2012 Winter;16(1):55-62. doi: 10.7812/TPP/11-134. PMID 22529761
- [Background] Munoz MA, Vila J, Cabanero M, Rebato C, Subirana I, Sala J, Marrugat J; ICAR (Intervencion en la Comunidad de Alto Riesgo cardiovascular) investigators. Efficacy of an intensive prevention program in coronary patients in primary care, a randomised clinical trial. Int J Cardiol. 2007 Jun 12;118(3):312-20. doi: 10.1016/j.ijcard.2006.07.015. Epub 2007 Jan 29. PMID 17261336
- [Background] Munoz MA, Rohlfs I, Masuet S, Rebato C, Cabanero M, Marrugat J; ICAR Study Group. Analysis of inequalities in secondary prevention of coronary heart disease in a universal coverage health care system. Eur J Public Health. 2006 Aug;16(4):361-7. doi: 10.1093/eurpub/cki202. Epub 2005 Oct 17. PMID 16230314
- [Background] Orozco-Beltran D, Brotons C, Moral I, Soriano N, Del Valle MA, Rodriguez AI, Pepio JM, Pastor A; investigadores del estudio PREseAP. [Factors affecting the control of blood pressure and lipid levels in patients with cardiovascular disease: the PREseAP Study]. Rev Esp Cardiol. 2008 Mar;61(3):317-21. Spanish. PMID 18361907
- [Background] Brotons C, Soriano N, Moral I, Rodrigo MP, Kloppe P, Rodriguez AI, Gonzalez ML, Arino D, Orozco D, Buitrago F, Pepio JM, Borras I; PREseAP study research team. Randomized clinical trial to assess the efficacy of a comprehensive programme of secondary prevention of cardiovascular disease in general practice: the PREseAP study. Rev Esp Cardiol. 2011 Jan;64(1):13-20. doi: 10.1016/j.recesp.2010.07.005. Epub 2010 Dec 30. PMID 21194823
- [Background] Murphy AW, Cupples ME, Smith SM, Byrne M, Byrne MC, Newell J; SPHERE study team. Effect of tailored practice and patient care plans on secondary prevention of heart disease in general practice: cluster randomised controlled trial. BMJ. 2009 Oct 29;339:b4220. doi: 10.1136/bmj.b4220. PMID 19875426
- [Background] Ortiz Tobarra MT, Orozco Beltran D, Gil Guillen V, Terol Molto C. [Frequency of attendance and degree of control of type-2 diabetic patients]. Aten Primaria. 2008 Mar;40(3):139-44. doi: 10.1157/13116629. Spanish. PMID 18373926
- [Background] Mira JJ, Orozco-Beltran D, Perez-Jover V, Martinez-Jimeno L, Gil-Guillen VF, Carratala-Munuera C, Sanchez-Molla M, Pertusa-Martinez S, Asencio-Aznar A. Physician patient communication failure facilitates medication errors in older polymedicated patients with multiple comorbidities. Fam Pract. 2013 Feb;30(1):56-63. doi: 10.1093/fampra/cms046. Epub 2012 Aug 17. PMID 22904014
- [Background] Marquez-Contreras E, de la Figuera-Von Wichmann M, Franch-Nadal J, Llisterri-Caro JL, Gil-Guillen V, Martin-de Pablos JL, Casado-Martinez JJ, Martell-Claros N. Do Patients With High Vascular Risk Take Antihypertensive Medication Correctly? Cumple-MEMS Study. Rev Esp Cardiol (Engl Ed). 2012 Jun;65(6):544-50. doi: 10.1016/j.recesp.2012.01.018. Epub 2012 Apr 19. PMID 22520867
- [Background] Gil-Guillen V, Orozco-Beltran D, Marquez-Contreras E, Durazo-Arvizu R, Cooper R, Pita-Fernandez S, Gonzalez-Segura D, Carratala-Munuera C, Martin de Pablo JL, Pallares V, Pertusa-Martinez S, Fernandez A, Redon J. Is there a predictive profile for clinical inertia in hypertensive patients? An observational, cross-sectional, multicentre study. Drugs Aging. 2011 Dec 1;28(12):981-92. doi: 10.2165/11596640-000000000-00000. PMID 22117096
- [Background] Gil-Guillen V, Orozco-Beltran D, Perez RP, Alfonso JL, Redon J, Pertusa-Martinez S, Navarro J, Cea-Calvo L, Quirce-Andres F, Merino-Sanchez J, Carratala C, Martin-Moreno JM. Clinical inertia in diagnosis and treatment of hypertension in primary care: quantification and associated factors. Blood Press. 2010 Feb;19(1):3-10. doi: 10.3109/08037050903350762. PMID 19929287
- [Background] Clark CE, Smith LF, Taylor RS, Campbell JL. Nurse-led interventions used to improve control of high blood pressure in people with diabetes: a systematic review and meta-analysis. Diabet Med. 2011 Mar;28(3):250-61. doi: 10.1111/j.1464-5491.2010.03204.x. PMID 21309833
- [Derived] Orozco-Beltran D, Ruescas-Escolano E, Navarro-Palazon AI, Cordero A, Gaubert-Tortosa M, Navarro-Perez J, Carratala-Munuera C, Pertusa-Martinez S, Soler-Bahilo E, Brotons-Munto F, Bort-Cubero J, Nunez-Martinez MA, Bertomeu-Martinez V, Gil-Guillen VF; PROPRESE research team. Effectiveness of a new health care organization model in primary care for chronic cardiovascular disease patients based on a multifactorial intervention: the PROPRESE randomized controlled trial. BMC Health Serv Res. 2013 Aug 2;13:293. doi: 10.1186/1472-6963-13-293. PMID 23915267